CLINICAL TRIAL: NCT01933841
Title: The Impact of Quantitative Neuromuscular Monitoring in the PACU on Residual Blockade and Postoperative Recovery
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Edward Sherwood, Professor, Vanderbilt University Medical Center
Other Study IDs: 131282
Record Dates: First submitted 2013-08-23; First posted 2013-09-02 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Muscle Weakness
Keywords: Post operative residual curarization; Neuromuscular blocking drugs
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Days 1-30: Adult surgery patients whose operations occurred during Days 1-30 after monitoring is introduced in the PACU. Patients will have their TOF ratio measured and recorded using a TOF-Watch SX. The nurse will monitor the patient and notify the provider of the patient's TOF-ratio if appropriate.
  Interventions: Device: TOF-Watch SX; Procedure: Notify the provider
- Days 31-60: Adult surgery patients whose operations occurred during Days 31-60 after monitoring is introduced in the PACU. Patients will have their TOF ratio measured and recorded using a TOF-Watch SX. The nurse will monitor the patient and notify the provider of the patient's TOF-ratio if appropriate.
  Interventions: Device: TOF-Watch SX; Procedure: Notify the provider
- Days 61-90: Adult surgery patients whose operations occurred during Days 61-90 after monitoring is introduced in the PACU. Patients will have their TOF ratio measured and recorded using a TOF-Watch SX. The nurse will monitor the patient and notify the provider of the patient's TOF-ratio if appropriate.
  Interventions: Device: TOF-Watch SX; Procedure: Notify the provider
- Days 91-120: Adult surgery patients whose operations occurred during Days 91-120 after monitoring is introduced in the PACU. Patients will have their TOF ratio measured and recorded using a TOF-Watch SX. The nurse will monitor the patient and notify the provider of the patient's TOF-ratio if appropriate.
  Interventions: Device: TOF-Watch SX; Procedure: Notify the provider

INTERVENTIONS:
Device: TOF-Watch SX — As part of standard care, patients who undergo intraoperative neuromuscular blockade will have their TOF ratio measured and recorded during their first 10 minutes in the PACU by perioperative nursing staff.
  Other Names: Acceleromyographic monitoring
Procedure: Notify the provider — Based on the TOF reading, the patient's PACU nurse will page the provider who administered the block and/or a designated "Reversal Support" team member. The page will identify the patient and notify the provider of the suboptimal TOF ratio.

SUMMARY:
Neuromuscular blocking drugs (NMBDs) provide anesthesiologists with powerful intraoperative tools, but their use carries the potential risk of serious postoperative complications. NMBD-induced muscle weakness that lingers into the postoperative period, known as postoperative residual curarization (PORC), is present in as many as 40% of all patients that receive neuromuscular blocking agents. The Post Anesthesia Care Unit will be introducing monitoring as part of standard of care. This study will collect data about patients who receive NMBDs and examine the impact of monitoring on incidences of PORC.

Our study is designed to test the following hypotheses:

Hypothesis 1: The initiation of quantitative TOF monitoring as part of the standard PACU entry evaluation will change practitioner behavior in a manner that decreases the incidence of PORC in surgical patients at VUMC.

Hypothesis 2: The initiation of the routine TOF monitoring program will decrease the incidence of short- and long-term postoperative complications at VUMC.

DETAILED DESCRIPTION:
Neuromuscular blocking drugs (NMBDs) provide anesthesiologists with powerful intraoperative tools, but their use carries the potential risk of serious postoperative complications. NMBD-induced muscle weakness that lingers into the postoperative period, known as postoperative residual curarization (PORC), is present in as many as 40% of all patients that receive neuromuscular blocking agents. Physiological data suggest that PORC impairs normal respiratory function, and compelling evidence suggests PORC impairs clinical recovery in the immediate postoperative period and prolongs PACU length of stay. However, despite the widespread use of NMBDs and the frequent occurrence of PORC, limitations in the literature prevent an understanding of their full impact on clinical outcomes. This study will collect data about patients who receive NMBDs and examine the impact of monitoring on incidences of PORC.

The incidence of PORC and postoperative complications after the introduction of monitoring in the PACU will be determined by measuring TOF ratios and tracking the postoperative outcomes in the surgical patients over time.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients > 18 years of age
* Received one or more NMBDs during surgery
* Surgery took place during the first 120 days following the introduction of TOF monitoring in the PACU

Exclusion Criteria:

* Surgical patients < 18 years of age
* Received no NMBDs during surgery
* Transfer from the OR to the PACU was delayed (by high PACU volume, for example)
* Had a procedure or has a preexisting condition that prevents accurate monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who receive an intraoperative neuromuscular blockade
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Decrease in incidence of postoperative residual curarization | 10 minute after arrival to PACU
  This aim will test the hypothesis that initiation of quantitative Train-Of-Four monitoring as part of the standard PACU entry evaluation will change practitioner behavior in a manner that decreases the incidence of PORC in surgical patients at Vanderbilt University Medical Center. Quantitative TOF monitoring will be introduced as a standard component of the PACU entry evaluation for all patients that receive NMBDs as part of their care. It is expected that the proportion of patients with TOF < 0.9 will decrease over time after initiation of the routine monitoring system.

SECONDARY OUTCOMES:
Decrease in the incidence of hemoglobin desaturation | PACU stay (Typically 1-2 hours post-operatively)
  This aim is part of a group of aims which will test the hypothesis that initiation of the routine TOF monitoring program will decrease short-term postoperative complications.
Decrease in need for reintubation | 24 hours after PACU entry
  This aim is part of a group of aims which will test the hypothesis that initiation of the routine TOF monitoring program will decrease short-term postoperative complications.
Decrease in length of stay in the PACU | PACU stay (Typically 1-2 hours post-operatively)
  This aim is part of a group of aims which will test the hypothesis that initiation of the routine TOF monitoring program will decrease short-term postoperative complications.
Decrease in incidence of perioperative pneumonia | 28 days post-operatively
  This aim is part of a group of aims which will test the hypothesis that initiation of the routine TOF monitoring program will decrease long-term postoperative complications.
Decrease in time to readiness for discharge | Hospital stay (Expected average of 3 days)
  This aim is part of a group of aims which will test the hypothesis that initiation of the routine TOF monitoring program will decrease long-term postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Edward R Sherwood, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No